CLINICAL TRIAL: NCT03203330
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center, Phase 3 Study to Determine the Efficacy of TG-C in Subjects With Kellgren and Lawrence Grade (KLG) 2 or 3 Osteoarthritis of the Knee
Brief Title: A Study to Determine the Safety and Efficacy of TG-C in Subjects With Kellgren and Lawrence Grade 2 or 3 OA of the Knee
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kolon TissueGene, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TGC-12301
Record Dates: First submitted 2017-06-21; First posted 2017-06-29 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Degenerative Osteoarthritis
Keywords: knee
MeSH Terms: conditions — Joint Diseases | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Treatment (TG-C) (Active Comparator): TG-C at 3 x 10e7 cells per single 2 mL intraarticular injection
  Interventions: Biological: TG-C
- Placebo Control (Normal Saline) (Placebo Comparator): Normal saline, single 2 mL intraarticular injection
  Interventions: Biological: Placebo Control

INTERVENTIONS:
Biological: TG-C — 2 mL injection of non-transduced human chondrocytes and irradiated transduced human GP2-293 cells expressing TGF-B1.
  Other Names: TissueGene-C
  Arms: Active Treatment (TG-C)
Biological: Placebo Control — 2 mL normal saline injection
  Other Names: Normal Saline
  Arms: Placebo Control (Normal Saline)

SUMMARY:
A randomized, double-blind, placebo-controlled, multi-center, phase 3 study to determine the safety and efficacy of TG-C in subjects with Kellgren and Lawrence Grade 2 or 3 Osteoarthritis of the Knee, Osteoarthritis Research Society International (OARSI) medial joint space narrowing (JSN) Grade 1 or 2 of the knee joint. TG-C is to be administered by a single intra-articular injection to the damaged joint area via ultrasound guidance. Patients will be followed for 24 months for safety and efficacy.

DETAILED DESCRIPTION:
This protocol is designed to assess the safety and efficacy of TG-C in treating symptoms of osteoarthritis of the knee and determining disease modifying effects of TG-C. This study is intended for the treatment of patients with KL Grade 2 and 3 osteoarthritis and OARSI JSN Grade 1 and 2. Assessments will be made on both the symptomatic effects of pain (VAS), function (WOMAC), and Quality of Life (SF-12) as well as the physical effects (JSW, MRI evaluations of whole knee joint organ tissues and structure) and biochemical biomarkers. This is a placebo-controlled study, TG-C will be compared to normal saline as a control. Additionally, this protocol is designed to evaluate the safety of TG-C. Safety will be evaluated by observation of the injection site for irritation or other effects, the incidence and severity of adverse events, and changes in physical examination findings, radiographic criteria, and laboratory tests. Patients will be followed for 24 months for both safety and efficacy with annual cancer surveillance questionnaires through 15 years post dosing for subjects who do not enroll in the Long Term Safety study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 or older
* BMI between 18.5 and 40
* KL Grade 2 or 3 knee OA
* OARSI Grade 1 or 2 medial JSN
* Pain >= 40 on VAS scale
* Written informed consent
* Using birth control

Exclusion Criteria:

* Knee symptoms that result in difficulty or inability to walk
* Knee effusion >2+
* Has Grade 3 OARSI JSN
* Has a score of 0 or >=5 on the cartilage feature of the WORMS at Screening
* MRI exam indicates fracture or tumor
* Has a positive result on RCR testing at Screening
* Has taken NSAIDS with 14 days of baseline
* Has taken steroidal anti-inflammatory medication within 2 months of baseline
* Chronic (>21 days) narcotic use
* Recent history (within 1 year) of drug or alcohol abuse
* Pregnant or lactating
* Has received injection to target knee within 2 months prior to study entry
* History of various disorders of the knee including but not limited to rheumatoid arthritis, psoriatic arthritis, autoimmune OA, chondrocalcinosis, gout, hemochromatosis, villonodular synovitis, or synovial chondromatosis
* Severe hip osteoarthritis ipsilateral to the target knee
* Ongoing infection disease including but not limited to HIV, Hepatitis B or C.
* Clinically significant congestive heart failure hepatic disease, kidney disease, adrenal insufficiency, acromegaly, uncontrolled hyper- or hypothyroidism, or non-specified uncontrolled endocrine disorder
* Uncontrolled diabetes based on a HbA1c > 8% at screening

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
Change in Knee Function as Assessed by the Western Ontario and McMaster Universities Index (WOMAC) | 12 months
  Assessment of change from baseline in target knee function using the WOMAC Osteoarthritis Index. The WOMAC is a proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee including pain, stiffness, and physical functioning of the joints. The response to the questions is in the form of a checked box associated with the response; None, Mild, Moderate, Severe and Extreme.
Change in Knee Pain as Assessed by VAS | 12 months
  Assessment of change from baseline in target knee pain using the Visual Analog Scale (VAS). The VAS is a method for the assessment of the intensity of pain. The VAS is a horizontal line, 100 mm in length and anchored by word descriptors at each end (no pain, very severe pain). The patient marks on the line at the point that represents their current state. The VAS score is determined by measuring in millimeters from the left hand end to the point of the mark. The score ranges from "0" or no pain to "100" very severe pain.

SECONDARY OUTCOMES:
MRI Assessment of Target Knee | 12 months
  Evaluation of the features of OA, as determined by structural changes of the knee joint, assessed by MRI
PCS of the SF-12 Questionnaire | 12 months
  Evaluation the Health-Related Quality of Life (HRQoL) as measured by the physical component score (PCS) of the 12-Item Short-Form Health Survey version 2 (SF-12v2®) questionnaire
WOMAC Total Score | 24 months
  Evaluation of the efficacy of TG-C with regard to knee function via WOMAC total score
Health Assessment Questionnaire Disability Index | 12 months
  Evaluation of the HRQoL as measured by the Health Assessment Questionnaire - Disability Index (HAQ-DI)

OTHER OUTCOMES:
Radiography for Structural Change in Knee Joint | Through 24 months
  Evaluate structural changes of the knee joint as determined by radiography (X-ray)
Efficacy of TG-C with Regard to Knee Function via WOMAC Total Score | At Months 3, 6, 9 and 18
  Evaluation of the efficacy of TG-C with regard to knee function via WOMAC total score
Efficacy of TG-C with Regard to Knee Function via WOMAC Pain, Function, and Stiffness Scores | Through 24 months
  Evaluate the efficacy of TG-C with regard to knee function via WOMAC® pain, function, and stiffness scores
Efficacy of TG-C with Regard to Knee Function via VAS Pain Score | At Day 1, Week 1, and Months 1, 3, 6, 9, 18 and 24
  Evaluation of the efficacy of TG-C with regard to knee function via VAS pain score at time points other than Month 12
OMERACT-OARSI Responder Analysis | 12 and 24 months
  Analysis of response using the Outcomes Measures in Rheumatoid Arthritis Clinical Trials (OMERACT)-OARSI responder criteria

CONTACTS AND LOCATIONS:
Overall Officials: Moon Jong Noh, PhD, Study Chair — Kolon TissueGene, Inc.
Locations (44):
- United States (44):
  - Jeffrey Davis, Birmingham, Alabama
  - Bradly Goodman, Birmingham, Alabama
  - Saima Chohan, Phoenix, Arizona
  - Nebojsa Skrepnik, Tucson, Arizona
  - Diraj Karnani, Apple Valley, California
  - Dan La, Covina, California
  - Scott Hacker, La Mesa, California
  - Eric Grigsby, Napa, California
  - Arthur Mabaquiao, San Diego, California
  - Timothy Davis, Santa Monica, California
  - Tien-I Su, Whittier, California
  - Mehul Desai, Washington D.C., District of Columbia
  - David Billmeier, Daytona Beach, Florida
  - Mercedes Ponce De Leon, Miami, Florida
  - Aurelio Torres-Consuegra, Miami, Florida
  - Edgar Gonzalez, Miami, Florida
  - Cathy Barnes, New Port Richey, Florida
  - Howard Chipman, Oldsmar, Florida
  - Richard Linn, Sunrise, Florida
  - Anand Patel, Winter Park, Florida
  - Sandeep Vaid, Newnan, Georgia
  - Dennis Levinson, Chicago, Illinois
  - Manish Jain, Chicago, Illinois
  - Hythem Shadid, Oak Brook, Illinois
  - Adil Fatakia, Marrero, Louisiana
  - James Nace, Baltimore, Maryland
  - Melvin Churchill, Lincoln, Nebraska
  - Jason Oh, New York, New York
  - Brett Gilbert, Durham, North Carolina
  - Jeremy Hoff, Wilmington, North Carolina
  - Yogesh Mittal, Tulsa, Oklahoma
  - Alan Kivitz, Duncansville, Pennsylvania
  - Edward Tavel, Columbia, South Carolina
  - Eric Loudermilk, Greenville, South Carolina
  - Harvey Bowles, Nashville, Tennessee
  - Daneshvari Solanki, Bellaire, Texas
  - Amr Morsy, Dallas, Texas
  - Haresh Boghara, DeSoto, Texas
  - Aldo Maspons, El Paso, Texas
  - Subodh Bhuchar, Houston, Texas
  - Brian MacGillivray, San Antonio, Texas
  - John Hemmersmeier, South Ogden, Utah
  - Kristen Holtz, Charlottesville, Virginia
  - Mark Hermann, Danville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mehta S, He T, Bajpayee AG. Recent advances in targeted drug delivery for treatment of osteoarthritis. Curr Opin Rheumatol. 2021 Jan;33(1):94-109. doi: 10.1097/BOR.0000000000000761. PMID 33229973